CLINICAL TRIAL: NCT06636279
Title: Clinical Effects of "Gas Bubble Technique" on Corneal Endothelial Recovery After Cataract Surgery
Brief Title: A Randomized Study of Gas Bubble Technique in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Rui Feng, PhD, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SichuanPPH2024331
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-04

CONDITIONS: Corneal Endothelial Damage Following the Hard Nuclear Cataract Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gas bubble group (Experimental): Inject the sterile air into the anterior chamber after the conventional cataract surgery to reduce the corneal endothelial damage
  Interventions: Procedure: Gas bubble technique
- The control group (No Intervention): Conventional cataract surgery

INTERVENTIONS:
Procedure: Gas bubble technique — Inject the sterile air into the anterior chamber after the conventional cataract surgery to reduce corneal endothelial damage
  Arms: Gas bubble group

SUMMARY:
To investigate the efficiency and safety of using "Gas Bubble Technique" to reduce corneal endothelial damage in hard nucleus cataract patients.

DETAILED DESCRIPTION:
The study is designed to: test the hypothesis that the "Gas Bubble Technique" is an effective method for reducing corneal endothelial damage. Describe and evaluate the effects of "Gas Bubble Technique" on a well-defined group of patients over a 1-month period following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent approved by the Ethics Committee
* 18-80 years of age
* Catract patients with hard nucleus (LOSIII N Score ≥4) who are scheduled for phacoemulsification
* Feasible for all visits and willing to follow instructions from the study investigator

Exclusion Criteria:

* Any ocular surgery history
* Currently diagnosis of severe ocular disease and under medication
* Uncontrolled systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Endothelial cell loss (ECL) | 1 week and 1 month
  The endothelial cell loss (ECL) was calculated as the percentage change in ECD from preoperative to postoperative values relative to the preoperative ECD.

SECONDARY OUTCOMES:
Central corneal thickness (CCT) increase rates | 1 week and 1 month
  CCT increase rates = ([postoperative CCT - preoperative CCT]/preoperative CCT) × 100%
Coefficient of variation (CV) | 1 week and 1 month
  Coefficient of variation reflected polymegathism
hexagonality (HEX) | 1 week and 1 month
  The percentage of hexagonality represented pleomorphism, indicating the ratio of hexagonal cells to cells of other shapes

OTHER OUTCOMES:
Intraocular pressure | 1day, 1week, 1 month
  Intraocular pressure measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
After the article is published, the data can be obtained from the corresponding author upon reasonable request